CLINICAL TRIAL: NCT00748683
Title: Development of an Integrated Health Care Environment for Elderly With RFID Technology
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Jin-Shin Lai, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20080816R
Record Dates: First submitted 2008-09-01; First posted 2008-09-08 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2008-09

CONDITIONS: Elderly
Keywords: elderly; longterm care
MeSH Terms: interventions — Radio Frequency Identification Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: RFID — A RFID tag attached on subjects' clothes 24hr a day during 1 month.

SUMMARY:
A falling prevention system will be established by RFID location and motion detection.

* Using RFID to detect participants' allocation indoor.
* Modifying environment parameters such as light, sound, to alert users if them enter a place with potential hazards.

Data exchange models will also developed in this project

* Interchanging different data including physiological data and RFID data into a database
* establishing interchange protocol according the HL7 standard

ELIGIBILITY:
Inclusion Criteria:

* Age above 65 year old
* Living in the Nursing home, Bei-Hu Branch, National Taiwan University Hospital
* with ability to independent ambulation (with or without assistive devices)

Exclusion Criteria:

* no ability to independent ambulation
* with infective diseases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Falling rate of participants | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shin Lai, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Nursing Home, Bei-Hu Branch, National Taiwan University Hospital, Taipei, Taiwan